CLINICAL TRIAL: NCT03071029
Title: Applying Behavioural Insights to Improve Take up of Post-abortion Family Planning: In-depth Study in Nepal
Brief Title: PAFP Provider Feedback Trial in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Stopes International (Other)
Collaborators: Ideas42 (Industry)
Responsible Party: Principal Investigator, Kathryn Church, Senior Scientific Advisor, Marie Stopes International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001-16
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Health Behavior
Keywords: family planning; reproductive health; abortion; health providers
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (receive data updates) (Experimental): Intervention clinics will receive a monthly poster that centres will receive which informs service providers of the PAFP LARC uptake rate at their centre. This is a step-wedged randomised controlled trial where all the clinics will eventually receive an intervention by the end of the study.
  Interventions: Behavioral: Monthly PAFP rates displayed at clinics.
- Control (no data updates) (No Intervention): Service providers at these clinics will not receive monthly information on PAFP LARC rates.

INTERVENTIONS:
Behavioral: Monthly PAFP rates displayed at clinics. — Providers will receive visual and text feedback on their centre's PAFP uptake rates as they compare to the uptake rates of other centres. The feedback will be delivered monthly in a physical paper format.
  Arms: Intervention (receive data updates)

SUMMARY:
A six-month RCT conducted within 36 health centres throughout urban and rural Nepal. The purpose of the RCT is to test the effectiveness of a peer comparison intervention at increasing uptake of long-acting reversible contraceptives (LARCs) as a percentage of PAFP uptake among clients who receive a safe abortion at a Marie Stopes International Nepal. The total sample size will be ~12,000 safe abortion clients. The primary outcome of interest is LARCs among safe abortion clients at Marie Stopes Centres in Nepal. The secondary outcome is to evaluate the impact of behaviorally designed intervention on the service providers' engagement in discussing measures to increase PAFP LARC uptake among women.

DETAILED DESCRIPTION:
The overall goal of the proposed research project is to increase uptake of long-acting reversible contraceptives (LARCs) among clients who receive a safe abortion at a Marie Stopes International - Nepal (MSI-N)/ Sunaulo Parivar Nepal (SPN) centre using a behaviourally-informed intervention: monthly feedback to service providers comparing their LARC uptake as a percentage of PAFP uptake performance to other centres. The impact of the intervention will be evaluated using a clustered, stepped wedge randomized controlled trial (RCT). The intervention will be implemented and data will be collected regularly from 36 centres over a period of 6 months. The RCT study design is stepped wedge, meaning that all health centres will begin in the control group and will be randomly assigned to begin receiving the treatment in 4 "steps". Each step will be 1 month in duration. The primary outcome of interest is LARC uptake as a percentage of PAFP uptake. The secondary outcome is type of method selected. The intervention consists of a monthly poster that centres will receive which shows service providers the PAFP LARC % performance at their centre as compared to 3 similar centres. The intervention was developed using a behavioral science methodology, including interviews with clients and service providers at 9 health centres and user-testing of the intervention with service providers at 4 health centres. Data used for this study will consist of daily PAFP LARC uptake data that is already being collected and consolidated at centres. The data will be securely shared between centres and the MSI-N central support office in Kathmandu on a weekly basis. Data will be securely shared between MSI-N and ideas monthly. Monitoring will consist of mystery client visits at each centre two times during the study period. At least one interview will be conducted with each service provider through the study period. The investigators will manually check 5% of all medical records to confirm that electronic data is accurate. Service providers will undergo written consent in order that they may choose to participate, or choose not to participate, in the study. Individual clients will be opted in to having their data shared for the purpose of the study. Clients will be notified about data sharing through posters and interactions with service providers and can choose not to have their data shared. All safe abortion clients, aged 18 and older, are eligible to have their data shared. Data from approximately 12,000 safe abortion clients will be required for the study. Strict confidentiality procedures in line with Marie Stopes International's best practices will be put into place to ensure that information made public or otherwise distributed outside the PIs and other key personnel cannot be linked to any individual client records. Results from the study will be published in a report, among other outputs, and the outcomes will be shared within MSI as well as with the wider sexual and reproductive health (SRH) community.

ELIGIBILITY:
Inclusion Criteria:

* All women over the age of 18 who receive safe abortion services at the 36 centres are eligible to participate in the study. Women will be opted in to the study.

Exclusion Criteria:

* Women <18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Long term reversible contraceptives uptake as a percentage of post-abortion family planning uptake among safe abortion clients within 2 weeks | 2 weeks post-abortion
  The study aims to observe a minimum 4% difference in PAFP LARC rates at two weeks post-abortion between intervention and control participants.

SECONDARY OUTCOMES:
Types of family planning method used after safe abortion procedure | 2 weeks post abortion
  % of participants using different types of family planning methods at two weeks post-abortion, including % using short-acting vs long-acting contraceptives.

CONTACTS AND LOCATIONS:
Overall Officials: Saugato Datta, Principal Investigator — Ideas42; Karina Lorenzana, Principal Investigator — Ideas42; Pragya Gartoulla, PhD, Principal Investigator — Marie Stopes Nepal
Locations (36):
- Nepal (36):
  - Marie Stopes Chuchchepati, Kathmandu, Bagati
  - Marie Stopes Gongabu, Kathmandu, Bagati
  - Marie Stopes Putalisadak, Kathmandu, Bagmati
  - Marie Stopes Satdobato, Kathmandu, Bagmati
  - Marie Stopes Banepa, Kavre, Bagmati
  - Marie Stopes Nuwakot, Nuwakot, Bagmati
  - Marie Stopes Kohalpur, Bānke, Bheri
  - Marie Stopes Surkhet, Surkhet, Bheri
  - Marie Stopes Parbat, Parbat, Dhaulagiri
  - Marie Stopes Gorkha, Gorkha, Gandaki
  - Marie Stopes Pokhara, Kāski̇̄, Gandaki
  - Marie Stopes Dumre, Tanahun, Gandaki
  - Marie Stopes Janakpur, Dhanusa, Janakpur
  - Marie Stopes Bardibas, Mahottari, Janakpur
  - Marie Stopes Lalbandi, Sarlahi, Janakpur
  - Marie Stopes Jumla, Jumla, Karnali
  - Marie Stopes Hile, Dhankutā, Koshi
  - Marie Stopes Biratnagar, Morang, Koshi
  - Marie Stopes Itahari, Sunsari, Koshi
  - Marie stopes Arghakhachi, Arghakhachi, Lumbini
  - Marie Stopes Gulmi, Gulmi, Lumbini
  - Marie Stopes Chandrauta, Kapilbastu, Lumbini
  - Marie Stopes Taulihawa, Kapilbastu, Lumbini
  - Marie Stopes Bhairahawa, Lumbini, Lumbini
  - Marie Stopes Butwal, Lumbini, Lumbini
  - Marie Stopes Bardghat, Nawalparasi, Lumbini
  - Marie Stopes Dadheldhura, Dadheldhura, Mahakali
  - Marie Stopes Ilam, Ilām, Mechi
  - Marie Stopes Birtamod, Jhapa, Mechi
  - Marie Stopes Narayanghat, Chitwan, Narayani
  - Marie Stopes Hetauda, Makwanpur, Narayani
  - Marie Stopes Birgunj, Parsa, Narayani
  - Marie Stopes Dang, Dāng, Rapti
  - Marie Stopes Pyuthan, Pyūthān, Rapti
  - Marie Stopes Lahan, Siraha, Sagarmatha
  - Marie Stopes Attariya clinic, Kailāli̇̄, Seti